CLINICAL TRIAL: NCT00317070
Title: A Randomized Controlled Trial to Evaluate the Efficacy and Tolerability of Intravesical Cocktail and Comparison With Intravesical Dimethyl Sulfoxide (DMSO) for the Treatment of Painful Bladder Syndrome Including Interstitial Cystitis (PBS/IC)
Brief Title: Trial Comparing Intravesical Cocktail With Intravesical Dimethyl Sulfoxide (DMSO) in Painful Bladder Syndrome/Interstitial Cystitis (PBS/IC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment, poor patient compliance, lack of funding
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Jerzy B Gajewski, Capital District Health Authority, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA010
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2008-05

CONDITIONS: Interstitial Cystitis; Bladder Diseases
Keywords: PBS/IC; Painful bladder syndrome including Interstitial cystitis
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Bladder Diseases | interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- DMSO (Active Comparator): Intravesical installation
  Interventions: Drug: dimethyl sulfoxide
- Cocktail (Experimental)
  Interventions: Drug: IC Cocktail

INTERVENTIONS:
Drug: dimethyl sulfoxide — intravesical installation 50 ml
  Arms: DMSO
Drug: IC Cocktail — * Heparin 10,000 units
  * Gentamicin 80 mg
  * Hydrocortisone sodium succinate (Solucortef) 100 mg
  * Lidocaine hydrochloride 1% 10 ml
  * Sodium Bicarbonate 8.4% 5 ml
  Arms: Cocktail

SUMMARY:
The primary objective of this study is to evaluate the efficacy and tolerability of the intravesical cocktail and its comparison with intravesical DMSO in a controlled trial for the treatment of painful bladder syndrome including interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants should be of age eighteen years or older
2. Participant has painful bladder syndrome and a score of 8 or greater on the painful bladder syndrome symptom index (O'Leary-Sant)
3. Participant should have frequency and urgency of micturition and bladder pain for at least 6 months
4. Participant should have voids at least 8 times during a 24 hour period and at least once during the night as documented in the voiding diary and questionnaire.
5. Urine culture should not show any evidence of urinary tract infection.
6. Participant should be able to understand, speak, and read English.
7. Participant should be willing to take part in the study, including signing this form after carefully reading it.
8. Participant consents to use a medically acceptable method of birth control throughout the entire study period and for four weeks after the study is completed. Medically acceptable methods of contraception that may be used by the study participants and/or their partners include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom and vaginal spermicide, surgical sterilization, vasectomy, or progestin implants or injections.
9. Failure of other treatments for PBS/IC like pentosan polysulfate (failure is defined as a score of +1 [slightly improved] or less on a global assessment response [GRA] 23 question to previous therapy)

Exclusion Criteria:

1. Participants who have undergone cystoscopy within 4 weeks of screening visit
2. Participants had other treatment given into the bladder in the past 4 weeks
3. Participants have used a new drug in the past 4 weeks which could affect bladder symptoms (some antidepressants, anticholinergics, antihistamines)
4. Past history of treatment with cyclophosphamide
5. A positive pregnancy test at the time of screening
6. Currently breast feeding
7. History of uterine, cervical, or vaginal cancer during the past 3 years
8. History of significant vaginitis
9. History of major surgery in the last 6 months
10. Positive tests for HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV)
11. History of immune deficiency diseases
12. History of bleeding disorders
13. History of serious social, mental, or medical conditions that would stop patient from taking part in the study
14. History of alcohol or drug abuse within the last 5 years
15. Participants who have history of prostate cancer or are being treated for chronic bacterial prostatitis
16. History of liver disease or significant medical problem which the investigator considers a risk for patient to be a part of the study
17. History of any of the following: neurogenic bladder radiation to pelvic area, inflammation of the bladder wall because of tuberculosis, schistosomiasis, bladder or ureteric calculi, or active genital herpes within 3 months of screening
18. Known hypersensitivity to one of the agents used in the intravesical instillation
19. Use of any investigational drug or device in the last 6 months
20. Participants who are unwilling or unable to abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
reduction of frequency of micturition | 16 weeks

SECONDARY OUTCOMES:
reduction in pain | 16 weeks
overall improvement of symptoms | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Gajewski, MD, FRCSC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Dept. of Urology, Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia, Canada